CLINICAL TRIAL: NCT00239837
Title: Preventing Problems for Girls in Foster Care
Brief Title: Prevention Program for Problem Behaviors in Girls in Foster Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Leslie D. Leve, Senior Fellow, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH054257 (NIH); R01MH054257 (NIH); R21DA027091 (NIH)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Juvenile Justice Involvement; Drug Abuse
Keywords: Adolescent; Foster Care; Female
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Middle School Success Intervention (MSS) (Experimental): Middle School Success Intervention (MSS): Participants receive the preventative intervention
  Interventions: Behavioral: Middle School Success Intervention (MSS)
- Foster Care Services as Usual (No Intervention): Foster Care Services as Usual: Participants continue with usual foster care

INTERVENTIONS:
Behavioral: Middle School Success Intervention (MSS) — This is a 10-month, psychosocial intervention for foster parents and girls, with administration of the intervention beginning the summer before entry into middle school. The intervention consists of: (1) six summer Pride groups for the girls, (2) six summer parenting intervention sessions for the foster parents; (3) weekly foster parent training and support sessions for foster parents during the first year of middle school; and (4) weekly individual skills training for the girls during the first year of middle school.
  Other Names: KEEP SAFE
  Arms: Middle School Success Intervention (MSS)

SUMMARY:
This study will determine the efficacy of a parent-involved intervention in preventing problem behavior in middle school girls who are currently in foster care.

DETAILED DESCRIPTION:
The transition from elementary school to middle school presents a complex set of challenges for adolescents. These include increased expectations for time management and self-monitoring, renegotiation of rules and boundaries with parents, increased peer influence, and pubertal changes. For children in foster care, this transition is further complicated by issues such as a possible history of maltreatment, unpredictable changes in their living situations, and difficulty explaining their foster care background to peers and teachers. Such issues may be more serious for girls in foster care. Social problems for these girls in middle school can lead to a number of negative effects, including delinquency, substance abuse, poor school performance, mental health problems, and participation in risky sexual behavior. Despite such risks, adolescent girls are less likely to receive specialty mental health or school-based services than their male counterparts. This study is aimed at determining the effectiveness of a preventive intervention for preadolescent girls living in foster/kinship care. The intervention targets include preventing delinquency, initiation of substance use, participation in risky sexual behavior, school truancy and failure, and mental health problems.

Participants were randomly assigned to receive either the preventive intervention or usual foster care services in the summer before entering middle school (typically sixth grade). The preventive intervention consisted of weekly training and support sessions for both participants and their foster or kin parents. The sessions began at study start and continued throughout participants' first year in middle school. Participants' relationship development, delinquency, school behavior and performance, sexual behavior, and substance use were assessed through questionnaires. Parenting practices were assessed through interviews. Assessments were conducted at study entry and at Months 6, 12, and 24, and 36. A new, follow-up assessment on the girls' decision making was conducted at age 14-16.

ELIGIBILITY:
Inclusion Criteria:

* Living in a foster home or receiving kinship care
* Are about to enter middle school
* Oregon resident
* Guardian willing to provide informed consent
* Female

Exclusion Criteria:

* male
* not in foster care
* not living in Oregon

Ages: 10 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2003-12; Primary Completion 2009-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Leve, PhD, Principal Investigator — University of Oregon
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

REFERENCES:
- [Background] Chamberlain P, Leve LD, Smith DK. Preventing Behavior Problems and Health-risking Behaviors in Girls in Foster Care. Int J Behav Consult Ther. 2006;2(4):518-530. doi: 10.1037/h0101004. PMID 18176629
- [Result] Mendle J, Leve LD, Van Ryzin M, Natsuaki MN, Ge X. Associations Between Early Life Stress, Child Maltreatment, and Pubertal Development Among Girls in Foster Care. J Res Adolesc. 2011 Dec 1;21(4):871-880. doi: 10.1111/j.1532-7795.2011.00746.x. PMID 22337616
- [Result] Natsuaki MN, Leve LD, Mendle J. Going through the rites of passage: timing and transition of menarche, childhood sexual abuse, and anxiety symptoms in girls. J Youth Adolesc. 2011 Oct;40(10):1357-70. doi: 10.1007/s10964-010-9622-6. Epub 2010 Dec 24. PMID 21184260
- [Result] Smith DK, Leve LD, Chamberlain P. Preventing internalizing and externalizing problems in girls in foster care as they enter middle school: impact of an intervention. Prev Sci. 2011 Sep;12(3):269-77. doi: 10.1007/s11121-011-0211-z. PMID 21475990
- [Result] Kim HK, Leve LD. Substance use and delinquency among middle school girls in foster care: a three-year follow-up of a randomized controlled trial. J Consult Clin Psychol. 2011 Dec;79(6):740-50. doi: 10.1037/a0025949. Epub 2011 Oct 17. PMID 22004305
- [Result] Mendle J, Leve LD, Van Ryzin M, Natsuaki MN. Linking Childhood Maltreatment with Girls' Internalizing Symptoms: Early Puberty as a Tipping Point. J Res Adolesc. 2014 Dec 1;24(4):689-702. doi: 10.1111/jora.12075. PMID 25419091
- [Result] Kim HK, Pears KC, Leve LD, Chamberlain PC, Smith DK. Intervention Effects on Health-Risking Sexual Behavior Among Girls in Foster Care: The Role of Placement Disruption and Tobacco and Marijuana Use. J Child Adolesc Subst Abuse. 2013 Nov 1;22(5):370-387. doi: 10.1080/1067828X.2013.788880. PMID 24043921
- [Result] Weller JA, Leve LD, Kim HK, Bhimji J, Fisher PA. Plasticity of risky decision making among maltreated adolescents: Evidence from a randomized controlled trial. Dev Psychopathol. 2015 May;27(2):535-51. doi: 10.1017/S0954579415000140. PMID 25997770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Child welfare staff members referred girls to the study between 2003-2006, by searching their database to gather information on all girls who were 10-12 years old, in their final year of elementary school, currently in foster care, and living in the targeted counties in Oregon.
Groups:
- 1 - Intervention: Participants receive the preventative intervention. The intervention consisted of two primary components: (a) six sessions of group-based caregiver management training for the foster parents and (b) six sessions of group-based skill-building sessions for the girls. The groups met twice a week for 3 weeks, with approximately seven participants in each group. The caregiver sessions were led by one facilitator and one cofacilitator. The girl sessions were led by one facilitator and three assistants to allow a high staff-to-girl ratio (1:2) for individualized attention, one-on-one modeling/practicing of new skills, and frequent reinforcement of positive behaviors. In addition to the summer group sessions, follow-up intervention services (i.e., ongoing training and support) were provided to the caregivers and girls in the intervention group once a week for 2 hr (foster parent meeting; one-on-one session for girls) during the first year of middle school.
- 2 - Foster Care Services as Usual: The girls and caregivers in the control condition received the usual services provided by the child welfare system, including services such as referrals to individual or family therapy, parenting classes for biological parents, and case monitoring. Of the girls in the control condition, 62% received individual counseling, 20% received family counseling, 22% received group counseling, 30% received mentoring, 37% received psychiatric support, and 40% received other counseling or therapy services (e.g., school counseling, academic support) during the first year of middle school. Note that many girls received more than one service, and therefore the percentages listed above exceed 100%. Child Welfare caseworkers managed each case and were responsible for making all decisions on referrals to community resources, including individual and family therapy and parenting classes.
Period: Overall Study
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Started | 48 | 52
6 Months | 48 | 50
Completed | 45 (3-year follow-up) | 45 (3-year follow-up)
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 52 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.48 (.51) | 11.59 (.45) | 11.54 (.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Delinquency
Description: 36 items from the general delinquency scale from the Self-Report Delinquency Scale (SRD; Elliott, Huizinga, & Ageton, 1985). Units on a scale. Girls were asked to rate how many times they had committed various delinquent acts (e.g., damaging or destroying properties, and stealing) in the past year, using an open-ended format. The mean of frequencies across these items was used to represent the level of delinquency for girls. The general delinquency scale scores ranged from 0 to 24 (full scale) and from 0 to 13 (log transformed). Higher scores indicate higher levels of delinquency.
Time Frame: Measured at Month 36
Population: FIML analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: log(units on a scale)
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
log(units on a scale) | .30 (.92) | .95 (2.69)

2. Secondary Outcome: Mental Health Problems
Description: Internalizing and externalizing symptoms at 12 and 24 months were measured with caregiver report on the Achenbach System of Empirically Based Assessment (ASEBA). This widely used checklist for psychopathological behaviors includes scales for behaviors such as Anxious/Depressed; Withdrawn; Somatic Complaints; Thought Problems; Attention Problems; Aggressive Behavior; Rule-Breaking Behavior; and Intrusive. The ASEBA has been shown to have both construct and content validity in the literature. For the present study, raw scores for the internalizing and externalizing symptoms subscales were used. Scores at 12 and 24 months were combined and averaged (mean). Units on a scale. Range = 0-66. Higher scores indicate higher levels of internalizing or externalizing problems.
Time Frame: Measured at Months 12 and 24
Population: Full information maximum likelihood (FIML) analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
units on a scale | 12.77 (8.53) | 12.50 (8.29)

3. Secondary Outcome: Participation in Risky Sexual Behaviors
Description: Eight items from the girls' in-person interviews were used to assess health risking sexual behavior at the 36-month followup. The girls reported on items such as touching a boy's body above or below the waist, having sexual intercourse, having sex with someone who they just met, or having sex with someone using drugs in the past 12 months. Positive answers to these items were totaled to represent the cumulative number of health-risking sexual behaviors. The frequency of the cumulative number of risky sexual acts ranged from 0 to 7. Units on a scale. Higher scores indicate more health-risking sexual behaviors.
Time Frame: Measured at Month 36
Population: FIML analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
units on a scale | .89 (1.17) | 1.69 (2.04)

4. Secondary Outcome: Social Competence
Description: Prosocial behavior was measured with a subscale from the Parent Daily Report (PDR; Chamberlain & Reid, 1987). The PDR was administered individually by telephone to foster parents on 3 consecutive or closely spaced days (1-3 days apart) at each assessment. A trained interviewer asked the foster parent whether a list of prosocial behaviors took place during the previous 24 hr (yes/no format). The prosocial scale was computed based on nine items, such as "cleans up after herself" and "do a favor for someone." The PDR was designed to avoid the potential bias of aggregate recall of frequency estimates. Studies have reported concurrent and predictive validity of the PDR checklist. The scores were averaged (mean) across calls from 3 days. Scores on prosocial behavior at 6 and 12 months were averaged and the mean across both time points was used in analysis. Units on a scale. Range = 0-9. Higher scores indicate more prosocial behavior.
Time Frame: Measured at Months 6, 12
Population: Full information maximum likelihood (FIML) analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
units on a scale | .80 (.12) | .74 (.14)

5. Secondary Outcome: Placement Changes
Description: Child welfare system records were collected at each assessment to determine the girls' placement changes (including the number and type of changes). Placement changes since the start of the study through 12 months were summed for each girl. The number of placement changes ranged from 0 to 7 during this period. Units on a scale. Higher scores indicate more placement changes.
Time Frame: Measured at Months 6 and 12
Population: Full information maximum likelihood (FIML) analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: placement changes
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
placement changes | .33 (1.05) | .76 (1.19)

6. Primary Outcome: Tobacco Use
Description: The girls were asked how many times in the past year they had smoked cigarettes or chewed tobacco. The response scale ranged from 1 (never) through 9 (daily). Units on a scale.
Time Frame: Measured at Month 36
Population: Full information maximum likelihood (FIML) analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: log(units on a scale)
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
log(units on a scale) | 1.49 (1.63) | 2.36 (2.49)

7. Primary Outcome: Marijuana Use
Description: The girls were asked how many times in the past year they had used marijuana. The response scale ranged from 1 (never) through 9 (daily). Units on a scale. Log transformed.
Time Frame: Measured at Month 36
Population: Full information maximum likelihood (FIML) analysis includes estimation of all cases even when missing data are present
Measure: Mean (Standard Deviation); unit: log(units on a scale)
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Number analyzed (Participants) | 48 | 52
log(units on a scale) | 1.29 (.82) | 2.33 (2.43)

8. Secondary Outcome: Decision Making
Description: "Cups" task (Weller et al., 2007). On each trial, participants see 2 arrays with equal number of X cups (2, 3, or 5) each. On gain trials, participants informed that under each cup in one array is 1 quarter, and the other array includes 1 cup with Y quarters (either 2, 3, or 5), but the other cups have 0 quarters. Choosing from the riskless side leads to a sure gain of 1 quarter while choosing the risky side can lead to gain of Y quarters or no quarters. On loss trials, participants shown that choosing cup from 1 array will lead to 1 quarter taken away while choosing cup from other array will lead to no quarters or Y quarters taken. Cups task consists of 54 trials of 3 trials each of all combinations of 2 levels of domain (gain, loss). Expected Value Sensitivity (EV) calculated by subtracting proportion of risky choices made when EV actually favored the sure choice from proportion of risky choices made on trials where EV favored risky option. Score can range from -1.0 to -1.0.
Time Frame: Measured at age 15-17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Middle School Success Intervention (MSS) | Foster Care Services as Usual
Number analyzed (Participants) | 45 | 47
units on a scale
  EV Sensitive in Loss Domain | .1383 (.22617) | .0378 (.18861)
  EV Sensitivity in Gain Domain | .2123 (.2282) | .2743 (.2429)
Statistical Analysis 1: Comparison: Middle School Success Intervention (MSS) vs Foster Care Services as Usual; Test type: Superiority or Other; p = .008, Regression, Logistic; Data analyzed using repeated logistic regression model (generalized estimating equations). Domain X EV Level X Group interaction tested; Wald χ2 = 7.14 — We began the analyses with a full-factorial model regressing choice on domain (gain=1, loss=0), the EV of the risky choice relative to the safe option (EV; range = -.38 to +.38), and dummy-coded treatment groups (Control= -1, Intervention =1)

ADVERSE EVENTS:
Arm/Group | 1 - Intervention | 2 - Foster Care Services as Usual
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 0/48 | 0/52

LIMITATIONS AND CAVEATS:
Sample is relatively small in size, and limited to girls in foster care in two Oregon Counties

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No